CLINICAL TRIAL: NCT01074242
Title: Re-examination Study for General Vaccine Use to Assess the Safety Profile of ROTATEQ in Usual Practice
Brief Title: ROTATEQ Reexamination Study (V260-037)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: V260-037; 2010_012 (Other: Merck)
Record Dates: First submitted 2010-02-22; First posted 2010-02-24 (Estimated); Results first posted 2014-03-27 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Gastroenteritis Rotavirus
Keywords: Gastroenteritis rotavirus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rotateq: Korean Infants vaccinated with Rotateq in usual practice. The Rotateq vaccination series consists of 3 ready-to-use liquid (oral) doses with the first dose to be administered at age 6-12 weeks and subsequent doses to be administered at 4 to 10-week intervals.

SUMMARY:
This survey is conducted for preparing application materials for re-examination under the Pharmaceutical Affairs Laws and its Enforcement Regulation, its aim is to reconfirm the clinical usefulness of Rotateq through collecting the safety information according to the Re-examination Regulation for New Drugs.

ELIGIBILITY:
Inclusion Criteria:

* Infants Who Are Vaccinated With Rotateq For The Prevention Of Rotavirus Gastroenteritis Within Local Labeling Will Be Included

Exclusion Criteria:

* Participants who are vaccinated with Rotateq before study start
* Participant who has a contraindication to Rotateq according to the local label

Ages: 6 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 6-32 week old Korean Infants who are vaccinated with Rotateq in usual practice
Sampling Method: Probability Sample
Enrollment: 3798 (Actual)
Dates: Start 2007-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/search.html?kw=V260-037

RESULTS

PARTICIPANT FLOW:
Groups:
- Rotateq: Korean infants vaccinated with Rotateq in usual practice
Period: Overall Study
Arm/Group | Rotateq
Started | 3798
Received at Least 1 Dose of Vaccine | 3395
Completed | 3395
Not Completed | 403
Not completed — Case report before date of contract | 40
Not completed — Lost to Follow-up | 1
Not completed — Case report unclear | 6
Not completed — Violation of vaccine dose or dosage | 351
Not completed — Duplicate Case Report Form | 5

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were reported for all enrolled participants who received at least 1 dose of study vaccine
Arm/Group | Rotateq
Number analyzed (Participants) | 3395
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 9.57 (1.03)
Age, Customized [Number; unit: Participants]
  <8 weeks | 90
  Between 8 and 10 weeks | 2740
  >10 weeks | 565
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1692
  Male | 1703

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Any Adverse Experience
Description: An adverse experience is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the product. Any worsening of a preexisting condition which is temporally associated with the use of the study vaccine is also an adverse experience.
Time Frame: Up to 42 days after any Rotateq vaccination
Population: All enrolled participants who received at least 1 dose of study vaccine were included in the analysis
Measure: Number; unit: Percent of participants
Arm/Group | Rotateq
Number analyzed (Participants) | 3395
Percent of participants | 22.12

2. Primary Outcome: Percentage of Participants With Any Adverse Drug Reaction
Description: An adverse drug reaction was an adverse experience for which a causal relationship to the study drug could not be ruled out
Time Frame: Up to 42 days after any Rotateq vaccination
Population: All enrolled participants who received at least 1 dose of study vaccine were included in the analysis
Measure: Number; unit: Percent of participants
Arm/Group | Rotateq
Number analyzed (Participants) | 3395
Percent of participants | 4.27

ADVERSE EVENTS:
Time Frame: Up to 42 days after any Rotateq vaccination
Description: All enrolled participants who received at least 1 dose of study vaccine were included in the analysis
Arm/Group | Rotateq
Serious Adverse Events (participants affected / at risk) | 8/3395
Other Adverse Events (participants affected / at risk) | 210/3395
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotateq (N=3395)
Gastroenteritis (Infections and infestations) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (4)
Urinary tract infection (Infections and infestations) | 3 (3)
Enteritis (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotateq (N=3395)
Nasopharyngitis (Infections and infestations) | 210 (263)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In regard to surveillance results, any publication should be agreed by the sponsor in advance